CLINICAL TRIAL: NCT05410314
Title: Nutritional Supplement Based on Myo-inositol-D-chiro-inositol: Effectiveness on the Reproductive System Functionality in Long-term Survivors of Lymphoma
Brief Title: Nutritional Supplement Based on Myo-inositol-D-chiro-inositoln in Long-term Survivors of Lymphoma
Acronym: Linf-inositol
Status: Completed | Type: Observational
Sponsor: University of Bari Aldo Moro (Other)
Responsible Party: Principal Investigator, MIRIAM DELLINO, UNIBA, University of Bari Aldo Moro
Other Study IDs: UNIBA
Record Dates: First submitted 2022-05-29; First posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-05

CONDITIONS: Lymphoma, Hodgkin; Menstrual Irregularity; Fertility Disorders
MeSH Terms: conditions — Hodgkin Disease; Menstruation Disturbances | interventions — Inositol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cHL (85%) and DLBCL (15%): Patients enrolled in this study are cHL (85%) and DLBCL (15%) long-term survivors, treated mainly with ABVD+ radiotherapy (not under diaphragmatic and pelvic irradiation), without relapse (during quinquennial follow-up) who are followed at the clinic dedicated to fertility in oncology of our Department, which is a regional referral center for this purpose. Therefore, the investigators conducted a prospective observational controlled study on two groups: the first one (A group) underwent oral supplementation with MIC for 12 months; the second group (B group) underwent follow-up without any nutritional supplement for 12 months
  Interventions: Drug: Myo-Inositol and D-Chiro-Inositol (MIC)

INTERVENTIONS:
Drug: Myo-Inositol and D-Chiro-Inositol (MIC) — Both groups were followed up for 12 months, in T0 (during first evaluation), and T12 (after twelve months) with blood test for AMH (ng/ml).

SUMMARY:
The progressive improvement of lymphoma treatment has led to an important prolongation of patient survival and life expectancy. Therefore, the principal International scientific societies of oncology, recommend Long-term Survivors of Lymphoma to join fertility programs. Specifically, fertile age patients should be assisted by a multi-disciplinary team including specialists dedicated to fertility preservation in oncology, in order to support the completion of the reproductive project. In general population, the use of Inositol was spready considered an effectives choice to contrast ovarian dysfunction with consequently improvement of reproductive outcomes, so it may represent an adjuvant strategy for this purpose. Therefore, the investigators conducted a pilot study to evaluate the potentialities of this nutritional supplement with the aim to optimize the reproductive function in Long-term Survivors of Lymphoma. Despite the limited number of cases and short observational time, this pilot investigation could represent a potential cornerstone for further insights, discussions, and applications

DETAILED DESCRIPTION:
Anticancer regimens are usually used to treat patients with lymphoproliferative neoplasms with a consequently transitory or permanent damage to their reproductive functionalities. Rates of gonadotoxicity of each chemotherapy could be modulated according to dose intensity, number of courses, and type of agent or combination. Classical Hodgkin lymphoma (cHL) and Diffuse Large B-cell lymphoma (DLBCL), including primary mediastinal Large B-cell Lymphoma (PMBL) have usually higher incidence in the 2nd or 3rd decade of life and presents cure rates of more than 75% 3,4 These histotypes need a poli-chemotherapy with ABVD (adriamycin, bleomycin, vinblastine, dacarbazine), which involves the association of alkylating and non-alkylating agents.

The autologous hemato-poietic stem cell transplant (ASCT) is needed in about the 10% of cHL and the 40% of DLBCL and has higher impact on fertility compared to ABVD 6. Therefore, both the chemotherapy (damaging the primordial follicle pool and then the ovarian reserve, OR) and the radiotherapy (exclusively secondary to under diaphragmatic and pelvic irradiation) could represent a risk of gonadotoxicity . In this scenario, data concerning fertility in cHL have been mainly evaluated by the German Hodgkin Study Group (GHSG) and the European Organization for Research and Treatment of Cancer (EORTC) through amenorrhea and anti-Mullerian hormone (AMH) evaluation. Indeed, amenorrhea has been used in numerous research to assess the gonadotoxicity of oncological treatment and reflect ovarian function . Furthermore, AMH could represent a gonadotoxicity marker, since it decreases during chemotherapy and could improve after the end of treatment, depending upon specific treatment schemes . Literature showed that after early-stage disease treatment (2 -4 cycle), more than 90% of patients reported a low gonadotoxic effect with a regular menstrual cycle after therapy (median recovery of 1 year). For advanced stage diseases (treated with 6 courses of ABVD) the gonadotoxic effect vary on base of patient's aged. Indeed, the complete AMH restoring during the 3-years follow-up period, was detected in all women under 35 years, and only 37% of older ones . Moreover, in a Cochrane meta-analysis, gonadotropin-releasing hormone agonist (GnRHa)seems to be effective in shielding the ovaries during chemotherapy, in terms of treatment-related premature ovarian failure, ovulation and menstruation recovery.

Beyond the ovarian suppression with GnRHa, there are several well-established procedures (oocyte cryopreservation, ovarian cortex cryopreservation for woman and sperm cryopreservation for men) that could prevent impact of these therapies in young patients. Therefore, considering the increased life expectation nowadays of Long-term Survivors of Lymphoma (patients in complete remission of the disease for more than 5 years) a fertility program with multi-disciplinary counselling is indicated. Particularly, in order to assess the damages upcoming after anticancer therapies on reproductive organs, international scientific societies such as the American Society for Reproductive Medicine (ASRM) (Ethics Committee of American Society for Reproductive Medicine, 2013), the American Society of Clinical Oncology (ASCO), the European Society for Medical Oncology (ESMO) as well as the International Society for Fertility Preservation (ISFP), strongly recommend a personalized and multidisciplinary counseling for each patient. In particular, the surveillance programs for the management of long-term lymphoma survivors should involve a team with onco-hematologists, radiotherapists, cardiologists, an endocrinologist, a psychologist, gynecologist, urologist and a nutritional biologist. The goal is to provide individualized therapeutic possibilities to restore endocrine function. Following these recommendations, an ambulatorial service dedicated to fertile patients with oncological disease was instituted in our Clinic of Gynecology Oncology, aiming to perform a careful assessment of the fertility state and support the reproductive project of those patients.

In these women,the investigators primarily estimated AMH, Follicle stimulating hormone (FSH), Luteinizing hormones (LH), 17β-estradiol ,in association to antral follicles count (AFC) assessed by ultrasonography during the cycle follicular phase. During this clinical evaluation, several patients often reported menstrual irregularities due to anovulatory cycles (50%), dysmenorrhea (20%) and abnormal uterine bleeding (30%).

Considering these elements, one of the potential therapeutic options could be considered the oral supplementation with Myo-Inositol and D-Chiro-Inositol (MIC). Indeed, MIC over the years has tiptoed to come alongside the classic pharmacological therapies, with robust compliance, safety, and effectiveness. MIC showed great potentiality to contrast ovarian dysfunction and optimize the reproductive function.

Therefore, the investigators conducted a prospective observational controlled study, with the aim to assess the effects of oral supplementation with MIC on ovarian function parameters in Long-term Survivors of Lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Classical Hodgkin lymphoma (cHL) and Diffuse Large B-cell lymphoma (DLBCL) long survival

Exclusion Criteria:

Ages: 25 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: From January 2020 to January 2021, 90 Long-term Survivors of Lymphoma female patients, average age 34 years (range 25-44) were considered eligible for the study. Each patient was informed about the procedures and signed informed consent before the surgery to allow data collection for research purposes.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2020-02-07 (Actual); Primary Completion 2021-02-07 (Actual); Study Completion 2021-12-07 (Actual)

PRIMARY OUTCOMES:
Number of Lymphoma long-term survivors treated with myo-inositol-D-chiro-inositol: evaluation of the results on the reproduction apparatus | 12 months
  The investigatirs conducted a prospective observational controlled study on two groups: the first one (A group) underwent oral supplementation with myo-inositol-D-chiro-inositol for 12 months; the second group (B group) underwent follow-up without any nutritional supplement for 12 months.Moreover, the investigators reported for each patient the menstrual frequency ( oligomenorrhea <25 days , normal flow 25-36 days , polymenorrhea >36 days), the duration of the cycle (short < 3 days, normal: 3-7 days , long >7 days), the amount of the menstrual cycle (poor <30 ml, normal 30-80 ml, >80 ml abundant) and dysmenorrhea and dyspareunia (visual analogue scale VAS pain scale = 1 -10).In addition, results of blood tests and clinical data about menstrual regularity and dysmenorrhea, were reported on the same database.In addition, results of blood tests and clinical data about menstrual regularity and dysmenorrhea, were reported on the same database.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS - Istituto Oncologico"Giovanni PaoloII", Bari, Italy

IPD SHARING:
Plan to Share IPD: No
From January 2020 to January 2021, 90 Long-term Survivors of Lymphoma female patients, average age 34 years (range 25-44) were considered eligible for the study.